CLINICAL TRIAL: NCT03077984
Title: Study on the Clinical Efficacy of Chinese Medicine Treatment of Sequelae of Apoplexy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tongsheng Su (Other)
Responsible Party: Sponsor-Investigator, Tongsheng Su, Professor, Shaanxi Hospital of Traditional Chinese Medicine
Organization: Shaanxi Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201507001-05
Record Dates: First submitted 2017-01-24; First posted 2017-03-13 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the cohort of Chinese medicine treatment (Experimental): The cohort of Chinese medicine treatment uses its comprehensive program of TCM on the basis of treatment with western medicine, including Chinese Herbs, acupuncture and acupoint application therapies.
  Interventions: Combination Product: Chinese medicine treatment
- the cohort of western medicine treatment (No Intervention): The cohort of Western medicine treatment refers to the treatment of cerebrovascular disease prevention and cure guideline of China-related programmes, including anti-platelet aggregation, blood pressure,blood glucose,Blood Lipids lowering therapies.

INTERVENTIONS:
Combination Product: Chinese medicine treatment — The cohort of Chinese medicine treatment uses its comprehensive program of TCM on the basis of treatment with western medicine, including Chinese Herbs, acupuncture and acupoint application therapies.
  Arms: the cohort of Chinese medicine treatment

SUMMARY:
This project is one multi-center, a prospective cohort study, based on 1660 cases of ischemic stroke patients with the treatment of 3 months, and 21 months of follow-up observation in order to clarify the advantages and characteristics of integrated treatment of traditional Chinese medicine sequela of apoplexy; With the formation of curative effect, to highlight the advantage of the programme of comprehensive treatment of apoplectic sequela in traditional Chinese medicine and its compound preparation; To form a active medical service mode of stroke chronic disease management processes, as well as modalities and mechanisms for the evaluation of the curative effect.

DETAILED DESCRIPTION:
There are more than 7 million stroke patients in China , about 2 million new cases of stroke patients each year, has become the national first cause of death, approximately 3/4 percent of survivors lost the ability to work due to apoplexy admitted to hospital 41.5% patients for recurrent patients. There is the legacy of somatic dysfunction in 80% of patients after stroke, The remaining 55.4% of the patients with mental disorders, The northwest region of China is a high incidence of "Stroke Belt" and the health care system in Northwest China is very weak, The "four high and one low" problem become more and more serious in the northwest, Therefore, clerify the advantages and characteristics of traditional Chinese medicine comprehensive treatment of sequelae of apoplexy. The formation of the active medical service model under the mode of stroke chronic disease management processes, and the evaluation of the curative effect and mechanism of paramount importance. In this paper 1660 cases of ischemic stroke patients with integrated traditional Chinese medicine therapy for 3 months, And 21-month follow-up observation To identify the traditional Chinese medicine comprehensive treatment to reduce mortality in patients with ischemic stroke recurrence rate, to improve the degree of disability of limbs after stroke and the effect of the main symptom of sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Patients in accordance with the criteria for the diagnosis of cerebral infarction.
* Functional Defects of Extremities1≤MRS≤5.
* Age between 18 and 75 years old (including 18 and 75), No gender limitation.
* Patients who agreed to participate in clinical trials and signed the informed consent form.
* Patients with stable vital signs after two weeks.

Exclusion Criteria:

* Patients with cerebral infarction at acute phase.
* Patients with cerebral infarction, transient ischemic attack, cerebral hemorrhage and cerebral arteritis.
* Patients with AF, ain tumor, brain trauma, brain parasite disease and rheumatic heart disease.
* Patients with bleeding or severe bleeding within 3 months.
* Patients with severe hepatitis, Kidneys, blood and the metabolic system diseases.
* Pisabilities and viewers with NIHSS prescribed by law.(Physical disabilities such as blind, deaf, dumb, mental disorder, mental disorder).
* Patients with history of alcohol and drug abuse, will reduce the possibility or make it hard into the Project Group according to the researchers' judgment.
* Allergic constitutions and drug sensitivities.
* Patients in other clinical trials or clinical trials of other drugs for more than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1660 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
recurrence rate of ischemic stroke | to observe the recurrence rate of ischemic stroke 1 year later
  In this paper 1660 cases of ischemic stroke patients with integrated traditional Chinese medicine therapy for 3 months, And 21-month follow-up observation To identify the traditional Chinese medicine comprehensive treatment to reduce mortality in patients with ischemic stroke recurrence rate, to improve the degree of disability of limbs after stroke and the effect of the main symptom of sequelae.
improve the degree of disability of limbs after ischemic stroke | to observe the degree of disability of limbs after ischemic stroke 2 year later
  In this paper 1660 cases of ischemic stroke patients with integrated traditional Chinese medicine therapy for 3 months, And 21-month follow-up observation To identify the traditional Chinese medicine comprehensive treatment to improve the degree of disability of limbs after stroke and the effect of the main symptom of sequelae.

IPD SHARING:
Plan to Share IPD: Yes